CLINICAL TRIAL: NCT06111755
Title: Evaluating Digital Health Interventions To Promote Smoking Cessation
Brief Title: Quit Smoking Text Message Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000035868; IA-1049344 (Other Grant/Funding Number: American Lung Association)
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmokefreeTXT (Active Comparator): Daily smokers for at least 6 months who report an interest in quitting will be randomized to receive the National Cancer Institute's SmokefreeTXT.
  Interventions: Other: SmokefreeTXT
- SmokefreeTXT + smartband (Experimental): Daily smokers for at least 6 months who report an interest in quitting will be randomized to receive the National Cancer Institute's SmokefreeTXT + smartband.
  Interventions: Other: SmokefreeTXT; Device: Smartband

INTERVENTIONS:
Other: SmokefreeTXT — National Cancer Institute's SmokefreeTXT is a text message quit smoking program available nationally. Users sign up and choose a target quit date that is within 2 weeks of their signup date. Users receive 3-5 text messages per day for up to 2 weeks pre-quit and 6 weeks post-quit. The quit date can be reset as often as needed by the user.
Device: Smartband — A smartband that will track smoking in real-time and ask the individual to confirm/deny smoking. Participants will be asked to wear the smartband during their waking hours and to charge it overnight.
  Arms: SmokefreeTXT + smartband

SUMMARY:
This project will address research gaps and advance the science of smoking cessation by conducting a randomized controlled trial of an evidence-based, population-level quit smoking text messaging program with or without a smartband.

DETAILED DESCRIPTION:
Aim 1 of this study is to test within-treatment effects for smoking cessation. The primary outcome will be biochemically (cotinine)-confirmed 7-day point-prevalence abstinence (PPA) at end of treatment (8 weeks). Secondary outcomes will be percent days smoke-free, time to relapse, and rated treatment satisfaction.

Aim 2 of this study is to explore sex/gender differences in treatment effects for smoking cessation. Given established sex/gender differences in smoking behavior and cessation,randomization will be stratified by sex/gender and we will measure effects of sex/gender on outcomes. Effect sizes will be estimated for smoking outcomes by sex.

Outcomes will be evaluated for those who complete enrollment, defined as those who complete study onboarding.

ELIGIBILITY:
Inclusion Criteria:

* daily smokers for at least 6 months
* report an interest in quitting smoking.

Exclusion Criteria:

* reporting being currently enrolled in another quit smoking program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with cotinine confirmed 7-day point-prevalence abstinence (PPA) at end of treatment (8 weeks) | 8 weeks
  7-day PPA at end of treatment with be confirmed via cotinine testing in saliva

SECONDARY OUTCOMES:
Change in cigarettes smoked per day | baseline, 4 weeks and 8 weeks
  Change in average number cigarettes smoked per day by self report
Percent days smoke-free | up to 8 weeks
  Percentage of smoke-free days by self report
Average number of days to relapse | 2 weeks post quit date
  Relapse is defined as 7 consecutive days of smoking after quitting and will be measured using self-report or smartband detection. This will be assessed after their quit date.
Treatment satisfaction assessed using the Mobile Application Rating Scale User version | up to 8 weeks
  This 20-item scale uses 5-point multiple choice ratings and has 6 subscales. Scores are reported as: 1) mean app quality, which is the mean score for the 4 subscales engagement, functionality, aesthetics, information quality; 2) mean of the app subjective quality subscale, and 3) mean of the perceived impact subscale. Higher scores indicate higher app quality, higher app subjective quality, and higher perceived impact. Mean scores range 1-5, with higher scores indicate higher app quality, higher app subjective quality, and higher perceived impact.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Garrison, PhD, Principal Investigator — Yale University
Locations (1):
- National online recruitment, New Haven, Connecticut, United States